CLINICAL TRIAL: NCT01238458
Title: Phase II Study for Amyloid Binding Imaging Study of [18F]AV-45 in Patients With Mild Cognitive Impairment, Alzheimer's Disease and Healthy Volunteers
Acronym: [18F]AV-45
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tzu-Chen Yen, Nuclear Medicine, Chang Gung Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 98-1852A
Record Dates: First submitted 2010-10-21; First posted 2010-11-10 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Alzheimer's Disease
Keywords: [18F]AV-45 PET amyloid binding imaging; Alzheimer's disease; mild cognitive impartment,
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- [18F]AV-45 PET amyloid binding imaging (Experimental)
  Interventions: Drug: [18F]AV-45 PET amyloid binding imaging

INTERVENTIONS:
Drug: [18F]AV-45 PET amyloid binding imaging — This study will recruit a total of 150 evaluable subjects (30 cognitively normal volunteers, and 60 MCI, and 60 AD, respectively) Each evaluable subject involved in this study must fulfill all the inclusion and exclusion criteria according the subject grouping.
  Safety measurement will be evaluated by medical history, vital signs, physical examinations, laboratory examinations and collecting of adverse events.

SUMMARY:
This study will recruit a total of 150 evaluable subjects (30 cognitively normal volunteers, and 60 MCI(Mild cognitive impairment), and 60 AD(Alzheimer's disease), respectively) Each evaluable subject involved in this study must fulfill all the inclusion and exclusion criteria according the subject grouping.

Safety measurement will be evaluated by medical history, vital signs, physical examinations, laboratory examinations and collecting of adverse events.

This study is expected to be completed in a period of 3 years.

DETAILED DESCRIPTION:
The primary objective of this protocol is to address the feasibility of clinical utilization of [18F]AV-45 in various neurodegenerative diseases. Specifically, we will expand the database of [18F]AV-45 PET imaging in Alzheimer's disease and MCI patients to refine the definition of a positive scan in patient with AD and MCI as compared to healthy control. Secondary, we will expand the safety database of [18F]AV-45 PET imaging. In addition, the image characteristics and prevalence of Aß positivity will be evaluated in different subsets of MCI and AD patients.

ELIGIBILITY:
Inclusion Criteria:

* Both genders ≥ 50 years old.
* Written and dated informed consent by self or by legal representative, to be obtained before any of the study procedures.
* 30 cognitively normal volunteers with no evidence of significant cognitive impairment by history and psychometrictesting (MMSE > 24).
* 60 subjects with a diagnosis of AD according to the NINCDS-ADRDA criteria.
* 60 subjects with a diagnosis of MCI

Exclusion Criteria:

1. Pregnant or becoming pregnant during the study (as documented by pregnancy testing at screening or at any date during the study according to the PI discretion) or current breast feeding.
2. Modified Hachinski ischemic score of >4 or those who meet the NINDS-AIREN criteria for vascular dementia.
3. Any subject who has a clinically significant abnormal laboratory values, and/or clinically significant or unstable medical or psychiatric illness.

   * Clinically significant hepatic, renal, pulmonary, metabolic, or endocrine disturbances, especially thyroid disease;
   * Current clinically significant cardiovascular disease. Clinically significant cardiovascular disease usually includes one or more of the following:

     * cardiac surgery or myocardial infarction within the last 6 months;
     * unstable angina
     * coronary artery disease that required a change in medication within the last 3 months
     * decompensated congestive heart failure
     * significant cardiac arrhythmia or conduction disturbance, particularly those resulting in atrial or ventricular fibrillation, or causing syncope, near syncope, or other alterations in mental status
     * severe mitral or aortic valvular disease
     * uncontrolled high blood pressure
     * congenital heart disease
     * clinically significant abnormal result on ECG, including but not limited to QTc>450 msec iii. Clinically significant infectious disease, including AIDS or HIV infection or active hepatitis B, active hepatitis C, HIV-1, or HIV-2
4. History of drug or alcohol abuse within the last year, or prior prolonged history of abuse.
5. Patients who have the evidence of neurodegenerative disorders other than AD, cognitive impairment resulting from trauma or brain damage, brain infarction, clinically significant psychiatric disease, epilepsy, are excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-11; Primary Completion 2011-11 (Actual); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
To expand the safety database of [18F]AV-45 PET imaging | one year
  To expand the database of [18F]AV-45 PET imaging in Alzheimer's disease and MCI patients to refine the definition of a positive scan in patient with AD and MCI as compared to healthy control.

SECONDARY OUTCOMES:
To expand the safety database of [18F]AV-45 PET imaging | two year
  To expand the safety database of [18F]AV-45 PET imaging Safety variables include adverse event count, lab parameters, vital signs, and ECG. Comparison will be generally made to baseline, as appropriate.
  To understand prevalence of Aß positivity in patients with MCI and AD. Images will be visually examined by a trained radiologist or nuclear medicine physician who is blinded to the subject diagnosis and will be reported as either Aβ positive (AD-like) or Aβ negative (not AD-like). The prevalence of Aß positivity in patients with MCI and AD will be recorded for comparison.